CLINICAL TRIAL: NCT02176226
Title: Artificial Intelligence in a Mobile Intervention for Depression and Anxiety (AIM)
Brief Title: IntelliCare: Artificial Intelligence in a Mobile Intervention for Depression and Anxiety (AIM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Mohr, Director, Center for Behavioral Intervention Technologies; Professor, Department of Preventive Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH100482-01-FTIC; R01MH100482-01 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder; Anxiety Disorders
Keywords: Major Depressive Disorder; Anxiety Disorders; Behavior Therapy; Technology Assisted; Mobile Phone; Cellular Phone; Smartphone; App
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 8-Week Single Arm Field Trial (Experimental): Use of IntelliCare program for 8 weeks.
  Interventions: Behavioral: IntelliCare

INTERVENTIONS:
Behavioral: IntelliCare — Behavioral interventions for depression and anxiety via a mobile phone application, IntelliCare.

SUMMARY:
This study will evaluate a Smartphone intervention for depression and anxiety that uses machine learning to tailor treatment for patients. The intervention, referred to as IntelliCare, delivers patient-specific treatment material and motivational messaging via a mobile phone, to help individuals with depression and/or anxiety. Information and data received from the patient will inform the tailored treatment approach through machine learning. The purpose of this study is to obtain preliminary information on the feasibility and effectiveness of IntelliCare in improving symptoms of depression and anxiety.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common mental disorder, with up to 10.3% of the population experiencing the disorder in a given 12-month period. The relationship between depression and anxiety has been well documented. Depression is a significant predictor of future anxiety, and anxiety is a significant predictor of future onset of depression. Indeed, studies find that more than 50% of all individuals with MDD also have a current anxiety disorder. Although effective treatments have been developed over the years to address depression and anxiety, the lack of personalization and inability to adapt to patient needs or preferences contributes to poor treatment adherence and outcomes.

We are developing an intelligent treatment system that uses state of the art machine learning approaches within a mobile intervention application to treat MDD and anxiety. Machine learning, a branch of artificial intelligence, focuses on the development of algorithms that automatically improve and evolve based on collected data. The intervention, called IntelliCare, uses a mobile application to continuously collect patient data and adapt intervention content and motivational messaging to create a highly tailored and user-responsive treatment system.

During the pilot study, 200 participants with Major Depression and/or Anxiety will use Intellicare apps for up to 8 weeks and may be invited to provide feedback about their experience at two follow-up time points: weeks 4 and 8. All participants will first undergo initial assessments that will include a telephone interview and a series of online questionnaires about their mood. Eligible participants will receive up to 8 weeks of access to the IntelliCare system, which consists of apps with lessons and tools designed to teach skills for mood management. It is suggested that participants utilize the mobile phone tools every day. Each week, participants will receive a brief motivational intervention from a coach. This coach will also be available to participants via email throughout the 8 week study. We will use data from the pilot study to examine whether IntelliCare is a feasible and effective intervention. Data collected will also be used to develop and evaluate machine learning methods which will be used in the subsequent AIM trials.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for clinically significant symptoms of depression or anxiety using self-report measures used in screening for depression, as well as interviewer administered measures to ensure symptoms are not transitory and have been present for at least two weeks.
* Is familiar with the use of mobile phones
* Has an Android phone and is willing download the IntelliCare apps on their own device
* Is able to speak and read English
* Is at least 19 years of age
* Is able to give informed consent

Exclusion Criteria:

* Has visual, hearing, voice, or motor impairment that would prevent completion of study and treatment procedures
* Has any psychiatric condition for which participation in a clinical trial of psychotherapy may be either inappropriate or dangerous (e.g., psychotic disorders, bipolar disorders, dissociative disorders, obsessive compulsive disorder, severe post traumatic stress disorder, etc.).
* Exhibits severe suicidality, including ideation, plan, and intent.
* Currently receiving psychotherapy or planning to receive psychotherapy during the 8 weeks of the study.
* Participants who have been on an antidepressant or anxiolytic medication with no dose changes for 2 weeks and do not intend to change the dose will be eligible. Those who have been on the antidepressant or anxiolytic for less than 2 weeks or intend to have their medication optimized will be asked to wait for screening until they meet the 2-week criterion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Mohr, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Interested parties can contact the PI. Data may be made available if proposed analyses are consistent with the IRB regulations and a Data Use Agreement is established

REFERENCES:
- [Derived] Rubanovich CK, Mohr DC, Schueller SM. Health App Use Among Individuals With Symptoms of Depression and Anxiety: A Survey Study With Thematic Coding. JMIR Ment Health. 2017 Jun 23;4(2):e22. doi: 10.2196/mental.7603. PMID 28645891
- [Derived] Mohr DC, Tomasino KN, Lattie EG, Palac HL, Kwasny MJ, Weingardt K, Karr CJ, Kaiser SM, Rossom RC, Bardsley LR, Caccamo L, Stiles-Shields C, Schueller SM. IntelliCare: An Eclectic, Skills-Based App Suite for the Treatment of Depression and Anxiety. J Med Internet Res. 2017 Jan 5;19(1):e10. doi: 10.2196/jmir.6645. PMID 28057609

RESULTS

PARTICIPANT FLOW:
Groups:
- 8-Week Single Arm Field Trial: Use of IntelliCare program for 8 weeks.
  IntelliCare: Behavioral interventions for depression and anxiety via a suite of mobile phone applications, IntelliCare.
Period: Overall Study
Arm/Group | 8-Week Single Arm Field Trial
Started | 105
Completed | 96
Not Completed | 9
Not completed — Lost to Follow-up | 3
Not completed — Withdrew prior to treatment | 6

BASELINE CHARACTERISTICS:
Arm/Group | 8-Week Single Arm Field Trial
Number analyzed (Participants) | 105
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [27 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 88
  More than one race | 1
  Unknown or Not Reported | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 35
  Married or domestic partner | 38
  Separated | 1
  Divorced | 13
  Widowed | 3
  Living with significant other | 15
Education [Count of Participants; unit: Participants]
  Some high school | 1
  Completed high school or GED | 4
  Some college | 20
  2-year college (Associate) | 16
  4-year college (BA, BS) | 37
  Master's degree | 22
  Doctoral degree | 4
  Professional degree (MD, JD) | 1
Employment status [Count of Participants; unit: Participants]
  Employed | 76
  Unemployed | 11
  Disability | 8
  Retired | 5
  Other | 5
Number of hours per week spent working [Median (Inter-Quartile Range); unit: hours per week spent working] | 40 [7 to 40]
Income, yearly household income [Median (Inter-Quartile Range); unit: USD] | 63,000 [30,000 to 100,000]
Income, yearly personal gross income [Median (Inter-Quartile Range); unit: USD] | 35,000 [15,000 to 58,000]
Treatment [Count of Participants; unit: Participants]
  Psychotherapy | 23
  Pharmacotherapy | 66
  None | 16
Recruitment Source [Count of Participants; unit: Participants]
  HealthPartners Healthcare system | 38
  Web or social media | 16
  ResearchMatch | 11
  Other | 40

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9) - Depression Severity Module
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome. Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe.
Time Frame: Baseline, Week 4, and Week 8
Population: Two participants missed week 4 assessment; and two participants missed week 8 assessment. This is why number analyzed in Week 4 row and Week 8 row differs from overall.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Single Arm Field Trial
Number analyzed (Participants) | 96
units on a scale
  Baseline | 12.5 (4.3)
  Week 4: number analyzed (Participants) | 94
  Week 4 | 8.4 (4.1)
  Week 8: number analyzed (Participants) | 94
  Week 8 | 6.4 (4.3)
Statistical Analysis 1: Comparison: 8-Week Single Arm Field Trial; Test type: Superiority; p < .001, t-test, 2 sided

2. Primary Outcome: GAD-7 (Generalized Anxiety Disorder Scale-7)
Description: The GAD-7 is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. GAD-7 total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome. Specifically, scores of 1-4 indicate minimal anxiety symptoms; 5-9 is mild anxiety symptoms; 10-14 is moderate anxiety symptoms; and 15-21 is severe anxiety symptoms.
Time Frame: Baseline, Week 4, and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Single Arm Field Trial
Number analyzed (Participants) | 96
units on a scale
  Baseline | 10.9 (4.5)
  Week 4: number analyzed (Participants) | 94
  Week 4 | 7.1 (3.9)
  Week 8: number analyzed (Participants) | 94
  Week 8 | 5.8 (4.0)
Statistical Analysis 1: Comparison: 8-Week Single Arm Field Trial; Test type: Superiority; p < .001, t-test, 2 sided

3. Secondary Outcome: Mean Number of Treatment App Use Sessions by Study Week
Time Frame: Weekly for Two Months
Population: Of the 99 participants who initiated the treatment, 96.0% (95/99) continued to use the apps at week 5 and 90.1% (90/99) continued through week 8.
Measure: Mean (Standard Deviation); unit: number of treatment app use sessions
Arm/Group | 8-Week Single Arm Field Trial
Number analyzed (Participants) | 98
number of treatment app use sessions
  Week 1 | 20.09 (15.63)
  Week 2: number analyzed (Participants) | 97
  Week 2 | 22.79 (16.76)
  Week 3: number analyzed (Participants) | 97
  Week 3 | 24.1 (20.21)
  Week 4: number analyzed (Participants) | 94
  Week 4 | 25.33 (20.68)
  Week 5: number analyzed (Participants) | 94
  Week 5 | 26.07 (20.41)
  Week 6: number analyzed (Participants) | 91
  Week 6 | 26.25 (23.66)
  Week 7: number analyzed (Participants) | 89
  Week 7 | 23.44 (22.27)
  Week 8: number analyzed (Participants) | 90
  Week 8 | 23.3 (25.57)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 8-Week Single Arm Field Trial
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Informed Consent Form (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT02176226/ICF_000.pdf